CLINICAL TRIAL: NCT00016081
Title: A Randomized Phase III Study To Evaluate The Safety And Efficacy Or Ribavirin Inhaled Solution In Preventing Progression Of Upper Respiratory Tract Respiratory Syncytial Virus (RSV) Infection To RSV Pneumonia In Blood And Bone Marrow Transplant (BMT) Recipients
Brief Title: Ribavirin Compared With Standard Care in Treating Patients With Respiratory Syncytial Virus Following Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: 1290.00; FHCRC-1290.00; NCI-G01-1939; CDR0000068593 (Registry Identifier: PDQ)
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Infection
Keywords: infection
MeSH Terms: conditions — Infections | interventions — Ribavirin

INTERVENTIONS:
Drug: ribavirin

SUMMARY:
RATIONALE: Antivirals such as ribavirin are used to treat infections caused by viruses. It is not yet known if ribavirin is more effective than standard therapy in preventing pneumonia in patients who have respiratory syncytial virus (RSV) infection following stem cell transplantation.

PURPOSE: Randomized phase III trial to compare the effectiveness of ribavirin with that of standard therapy in preventing pneumonia in patients who have RSV infection following stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of aerosolized ribavirin vs standard supportive therapy, in terms of preventing progression of upper respiratory tract respiratory syncytial virus (RSV) infection to pneumonia, in patients with RSV following stem cell transplantation.
* Determine the safety of aerosolized ribavirin in this patient population.

OUTLINE: This is a randomized, investigator-blind, controlled, multicenter study. Patients are stratified according to engraftment status (pre vs post) and transplant type (HLA matched-related allogeneic, syngeneic, or autologous vs HLA mismatched-related or unrelated allogeneic). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive standard supportive care for immunocompromised patients with upper respiratory tract infections. Patient also receive aerosolized ribavirin by face mask, mist, or oxygen tent over 2 hours 3 times daily on days 1-10.
* Arm II: Patients receive standard supportive care as in arm I. Treatment continues in the absence of progression to pneumonia or unacceptable toxicity.

Patients are followed at days 14 and 28.

PROJECTED ACCRUAL: A total of 90 patients (45 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed upper respiratory tract respiratory syncytial virus (RSV) infection documented in nasopharyngeal-throat specimen by rapid antigen test (ELISA), IFA, or shell vial)

  * Signs or symptoms of upper respiratory tract infection (e.g., rhinorrhea and/or low-grade fever (under 101 degrees F with or without evidence of a sore throat)
* Received prior stem cell transplantation (SCT) and meet one of the following criteria:

  * Between start of conditioning (preparative) regimen and day 90 after allogeneic, autologous, or syngeneic SCT
  * Between days 91 and 180 after unrelated or HLA mismatch-related allogeneic SCT
  * Between days 91 and 180 after SCT with graft-versus-host disease requiring systemic steroids expected to continue throughout study
* No radiographic evidence of pneumonia

PATIENT CHARACTERISTICS:

Age:

* 2 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Pulmonary:

* Oxygen saturation 92-100% by pulse oximeter
* Normal respiratory rate for age

Other:

* No prior adverse reactions to ribavirin
* No clinical status that would preclude study
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior immunotherapy for RSV
* No prior or concurrent RSV hyperimmune globulin or monoclonal antibodies

Chemotherapy:

* Not specified

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior antiviral drugs with anti-RSV activity
* Bronchodilator treatment allowed for patients with asthma or a history of reactive airway disease and/or who develop bronchospasm
* Concurrent ganciclovir, foscarnet, or IV immunoglobulin allowed
* No mechanical ventilation
* No other concurrent anti-viral drugs with anti-RSV activity

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-03; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boeckh, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (4):
- United States (4):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Siteman Cancer Center, St Louis, Missouri
  - Fred Hutchinson Cancer Research Center, Seattle, Washington